CLINICAL TRIAL: NCT04595383
Title: Efficacy of an Electronic Communication Platform to Activate Diabetic Patients Treated With Insulin
Brief Title: Electronic Platform for Diabetic Patients Activation
Acronym: INSULINCOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Domingo Orozco, Principal investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/09
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Hypoglycemia; Hypoglycemia Acute
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care and usual communication with health professional
- Intervention (Experimental): They will be trained to use the ti.care platform and will be able to use it as a communication channel for any questions or clarification they require during the time elapsed between routine control visits. This platform will be a complement to the visits, but in no case will it replace them or be used as a diagnostic or therapeutic method. The platform does not have any treatment algorithm and only aims to facilitate communication between the patient at home and the health professional, both the doctor and the nurse educator. It will be used in a preventive and advisory manner for the patient for follow-up. In no case it will be used for emergencies. Daily during working hours from Monday to Friday, health professionals will review patient requests and respond to them.
  Interventions: Device: ti.care

INTERVENTIONS:
Device: ti.care — Electronic platform for doctor-patient communication
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the efficacy of an electronic platform for doctor-patient communication in order to reduce severe and non-severe hypoglycemia events as well as inadvertent hypoglycemia events.

DETAILED DESCRIPTION:
This is an open randomized clinical trial without drugs. Patients with type 2 diabetes and treated with insulin will be included. Patients allocated in the intervention group will use the electronic platform as a communication channel with their health provider during the time between visits.

The name of the platform is ti.care (https://ti.care/es) and it will be a complement of the control visits to resolve doubts through chats, email or video call. Health providers will answer the patient requests.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 17 years
* Patients with type 2 diabetes diagnosis
* Patients who start insulin treatment or with intensification of treatment
* Patients who sign informed consent

Exclusion Criteria:

* Patients with type 1 diabetes diagnosis
* Life expectancy less than one year
* Pregnancy
* Patients with dementia
* Patients with treatment different to insulin
* Patients who, in the opinion of the researcher, cannot follow the recommendations of the self-care health education plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from HbA1c level at 3 months | Baseline and at 3 months
  Change from HbA1c level at 3 months
Change from basal capillary blood glucose at 3 months | Baseline and at 3 months
  Change from basal capillary blood glucose at 3 months
Change from postprandial blood glucose at 3 months | Baseline and at 3 months
  Change from postprandial blood glucose at 3 months
Change from nocturnal blood glucose at 3 months | Baseline and at 3 months
  Change from nocturnal blood glucose at 3 months
Total hypoglycemia | At 3 months
  Number of total hypoglycemia events
Number of nocturnal hypoglycemia events | At 3 months
  Number of nocturnal hypoglycemia events
Number of inadvertent hypoglycemia events | At 3 months
  Number of inadvertent hypoglycemia events